CLINICAL TRIAL: NCT07204977
Title: Acamprosate in C9orf72 Hexanucleotide Repeat Expansion Amyotrophic Lateral Sclerosis (ACALS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002127; 002127-N
Record Dates: First submitted 2025-10-02; First posted 2025-10-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Clinical Trial; Acamprosate; C9ORF72
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Frontotemporal Dementia With Motor Neuron Disease | interventions — Acamprosate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): This is a single arm study, capturing the safety profile of acamprosate over the course of the study.
  Interventions: Drug: Acamprosate calcium

INTERVENTIONS:
Drug: Acamprosate calcium — tablet

SUMMARY:
Background:

Amyotrophic lateral sclerosis (ALS) is a disorder that damages nerve cells in the brain and spinal cord. It can cause muscle weakness, paralysis, and loss of movement. The symptoms grow worse over time. Half of all people with ALS live only 3 to 5 years after diagnosis. Current drug treatments can slow the progress of the disease, but they cannot stop or reverse it.

Objective:

To test a study drug (acamprosate) in people with ALS with a mutation in the C9orf72 gene.

Eligibility:

People aged 18 years and older with ALS. They must have a mutation in the C9orf72 gene.

Design:

Participants will have 13 visits over 32 weeks. Five visits will be at the clinic, and 8 visits will be by phone.

Participants will have a baseline visit of up to 3 days. They will have a physical exam with blood tests. They will have imaging scans and tests of their breathing ability. Their memory, thinking, and behavior will be assessed. They will have a neurologic exam to check their reflexes, strength, balance, eyes, and coordination. They will complete questionnaires about their daily life. They will have a lumbar puncture to collect fluid from the area around the spinal cord.

Acamprosate is a pill taken by mouth. Participants will take 2 pills by mouth 3 times a day with meals for 24 weeks. They will record their doses and any missed doses in a diary.

Baseline tests will be repeated during follow-up clinic visits. These tests may be spread out over 3 days.

During phone visits, participants will talk about how they are doing. They will review their diary with researchers.

DETAILED DESCRIPTION:
Study Description:

This study will evaluate the safety and clinical effects of acamprosate in patients diagnosed with amyotrophic lateral sclerosis who have a hexanucleotide repeat expansion in the C9orf72 gene. A drug repurposing evaluation using genomic data from C9orf72 genetic mutation carriers showed that acamprosate may have a neuroprotective effect in this group of patients in silico and experiments. To examine the in vitro effect, iPSC derived motor neurons from ALS patients with C9orf72 repeat expansion were treated with acamprosate and reduced cell death was observed. Exploratory endpoints will include the effect of acamprosate on ALS disease progression.

Objectives:

Primary objective: To assess the safety of acamprosate in patients with ALS and mutation in C9orf72.

Secondary objective: To investigate the clinical effects of acamprosate in patients with ALS and mutation in C9orf72.

Exploratory objective: To investigate the clinical, laboratory, and neuroimaging effects of acamprosate in patients with ALS and mutation in C9orf72.

Endpoints:

Primary endpoint: Adverse events (AEs), Serious Adverse Events (SAEs), and laboratory abnormalities during treatment. Each AE will be categorized according to its severity, its relation to the study intervention, its frequency, and its outcome.

Secondary endpoint: The change in ALS Functional Rating Scale-Revised (ALSFRS-R) score from baseline at predetermined time points during the study.

Exploratory endpoint: The change ALS disease severity and quality of life scales, neurodegeneration biomarkers, and neuroimaging measures from baseline at predetermined time points during the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following inclusion criteria:

1. Aged 18 years or older at the time of the screening visit.
2. Able to provide informed consent and comply with study procedures and availability for the duration of the study. If a participant lacks capacity to give consent, a Legally Authorized Representative (LAR) will be authorized to give consent on behalf of the individual.
3. Diagnosis of ALS (possible, probable, or definite according to the World Federation of Neurology El Escorial revised criteria or the Gold Coast Criteria) with or without mild cognitive impairment, mild behavioral impairment, or frontotemporal dementia (FTD).
4. CLIA-certified genetic testing showing a pathogenic hexanucleotide repeat expansion in the C9orf72 gene.
5. Symptom duration less than 2 years, or if greater than 2 years, disease progression at a rate that, in the judgement of the investigator, would allow for completion of the study.
6. If taking riluzole, edaravone, or phenylbutyrate/TUDCA, the participant must be on a stable dose for at least 30 days prior to the screening visit, or have stopped taking riluzole, edaravone, or phenylbutyrate/TUDCA at least 30 days prior to the baseline visit.
7. Participant must be competent to self-administer the medication as deemed by study team. Alternatively, participant must have a competent caregiver who can and will be responsible for administering the study drug. If there is no caregiver, another qualified individual must be available to administer the study drug.
8. Participant has established care with a neurologist and will maintain this clinical care throughout the study.
9. For females of reproductive potential: use of effective or highly effective contraception for at least one month prior to screening and agreement to use such a method during study participation and for an additional 8 weeks after the end of acamprosate administration. Participants of childbearing potential must have a negative pregnancy test at screening.
10. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Dependence on daytime mechanical ventilation (invasive or non-invasive, including Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPAP) at the time of the screening visit.
2. Participation in any other investigational drug trial or using investigational drug(s) (within 4 weeks prior to the Day 0 visit and thereafter).
3. Participants must not become pregnant or breastfeed for the duration of the study. Participants of childbearing potential must have a negative pregnancy test at screening and be non-lactating.
4. Men who are trying to become fathers or donate sperm.
5. History of positive test or positive result at screening for HIV.
6. History of severe sulfonamide allergy (i.e., anaphylaxis).
7. Presence of any of the following clinical conditions at the time of screening:

   1. Active drug abuse or alcoholism.
   2. Unstable medical condition that, in the opinion of the investigators, makes participation unsafe.
   3. Renal impairment estimated glomerular filtration rate <=60mg/dl or a creatinine clearance rate <= 50 milliliters per minute.
   4. Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days of the screening visit.
8. Safety Laboratory Criteria at the screening visit:

   1. Estimated glomerular filtration rate <=60mg/dl.
   2. Platelet concentration of <100,000/microl.
   3. PT and PTT >1.2 times the upper limit of normal.
   4. Hemoglobin <10mg/dL.
   5. Positive Hepatitis B Surface Antigen and Hepatitis C Virus Antibody
9. Participants who are unable to swallow tablets whole, as required by the administration guidelines. This includes individuals with any medical condition or physical limitation that impedes their ability to swallow solid dosage forms.
10. Participants who are dependent on a gastrostomy tube for medication administration. Since acamprosate is in tablet form that cannot be crushed or altered, it is unsuitable for administration through a gastrostomy tube.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety of acamprosate in patients with ALS and mutation in C9orf72. | Six months
  Incidence of adverse events and serious adverse events and abnormalities in laboratory tests (complete blood count, acute care panel, hepatic and mineral panel).

SECONDARY OUTCOMES:
To investigate the clinical effects of acamprosate in patients with ALS and mutation in C9orf72. | Six months.
  Total score on the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Y Kwan, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002127-N.html